CLINICAL TRIAL: NCT04733742
Title: Intravenous rhTNK-tPA Bridging With Endovascular Treatment Versus Endovascular Treatment Alone For Stroke Patient With Large Vessel Occlusion: A Multicenter, Randomized Controlled Trial
Brief Title: Endovascular Treatment With Versus Without Intravenous rhTNK-tPA in Stroke
Acronym: BRIDGE-TNK
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Xinqiao Hospital of Chongqing (Other)
Collaborators: CSPC RECOMGEN PHARMACEUTICAL (GUANGZHOU) CO.,LTD (Unknown)
Responsible Party: Principal Investigator, Zhongming Qiu, Professor, Xinqiao Hospital of Chongqing
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BRIDGE-TNK
Record Dates: First submitted 2021-01-26; First posted 2021-02-02 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Stroke, Acute; Stroke, Ischemic
Keywords: Thrombolysis; Endovascular treatment; rhTNK-tPA
MeSH Terms: conditions — Stroke; Ischemic Stroke | interventions — Tenecteplase; TNK-tissue plasminogen activator

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conbined treatment group (Experimental): intravenous tenecteplase bridging with endovascular treatment
  Interventions: Drug: rhTNK-tPA; Other: Endovascular treatment
- Endovascular treatment alone group (Active Comparator): endovascular treatment alone
  Interventions: Other: Endovascular treatment

INTERVENTIONS:
Drug: rhTNK-tPA — intravenous thrombolysis with rhTNK-tPA followed by endovascular treatment
  Other Names: TNKase; TNK-tPA
  Arms: Conbined treatment group
Other: Endovascular treatment — endovascular treatment
  Other Names: intra-arterial treatment; interventional therapy

SUMMARY:
The purpose of this trial is to investigate whether intravenous rhTNK-tPA prior to endovascular treatment can improve 90-day functional outcome of stroke patients with large vessel occlusion who are thrombolysis-eligible within 4.5 hours of symptom onset.

DETAILED DESCRIPTION:
The DEVT, SKIP and DIRECT-MT trials showed that endovascular treatment alone is not inferior to intravenous alteplase bridging with endovascular treatment in terms of achieving 90-day functional independence for stroke patients with large vessel occlusion. The EXTEND-IA TNK part 1 and part 2 demonstrated that intravenous thrombolysis with tenecteplase is superior to alteplase before endovascular treatment. However, it is unclear whether intravenous tenecteplase bridging with endovascular treatment is superior to endovascular treatment alone. The purpose of this trial is to investigate whether intravenous rhTNK-tPA bridging with endovascular treatment is better than endovascular treatment alone for stroke patients with large vessel occlusion who are thrombolysis-eligible within 4.5 hours of onset.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older;
2. Patient with acute ischemic stroke who is eligible for intravenous thrombolysis treatment within 4.5 hours of time last known well;
3. No significant prestroke functional disability: for age <80 years, prestroke modified Rankin scale (mRS) ≤2; for age ≥80 years, prestroke mRS ≤1;
4. MCA-M1 or -M2, basilar artery, or posterior cerebral artery-P1 occlusion proved by CTA/MRA;
5. EVT is planned by clinical care team;
6. Written informed consent is obtained from patients and/or their legal representatives.

Exclusion Criteria:

1. Intracranial hemorrhage on baseline CT or MR
2. Contraindication to intravenous thrombolytics
3. Already received intravenous thrombolytic after index stroke
4. Known pregnancy, or breastfeeding, or serum beta human chorionic gonadotropin test is positive on admission
5. Contraindication to radiographic contrast agents, nickel, titanium metals or their alloys
6. Current participation in another investigational drug clinical trial
7. Arterial tortuosity and/or other arterial disease that would lead to unstable access platform or prevent the thrombectomy device from reaching the target vessel
8. Patient with a preexisting neurological or psychiatric disease that would confound the outcome assessments
9. Patient with occlusions in two or more vascular territories (e.g. bilateral territories, or anterior and posterior circulation)
10. Mass effect or intracranial neoplasm on baseline CT or MR (except small meningioma)
11. Intracranial arteriovenous malformation or aneurysm on baseline CT or MR angiography
12. Any terminal disease with a life expectancy less than half a year
13. Unlikely to be available for follow-up at 90 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Actual)
Dates: Start 2022-05-09 (Actual); Primary Completion 2024-12-16 (Actual); Study Completion 2025-02-07 (Actual)

PRIMARY OUTCOMES:
Proportion of patients functionally independent (mRS score 0 to 2) at 90 days | 90 days
  functional independence

SECONDARY OUTCOMES:
Substantial reperfusion at initial angiogram | within 5 minutes at initial angiogram
  evaluate effect of tenecteplase on reperfusion
Successful reperfusion at end-of-procedure angiography | 15 minutes after initial angiogram
  evaluate vascular patency after thrombectomy
First-pass reperfusion | After artery puncture, but before thrombectomy
  defined as Expanded Treatment in Cerebral Infarction ≥2c after the first thrombectomy pass
Modified first-pass reperfusion | After artery puncture, but before thrombectomy
  defined as Expanded Treatment in Cerebral Infarction ≥2b after the first thrombectomy pass
National Institutes of Health Stroke Scale (NIHSS) score | 5 to 7 days or discharge
  Neurological status
modified Rankin scale score | 90 days
  disability level
Proportion of patients non-disabled (mRS score 0 to 1) or return to pre-morbid mRS score at 90 days (for patients with mRS > 1) | 90 days
  excellent outcome
Proportion of patients ambulatory or bodily needs-capable or better (mRS score 0 to 3) | 90 days
  ambulatory or bodily needs-capable or better
Health-related quality of life, assessed with the European Quality Five Dimensions Five Level scale (EQ-5D-5L) | 90 days
  Health-related quality of life
Any radiologic intracranial hemorrhage within 48 hours | within 48 hours after endovascular treatment
  evaluate intracranial hemorrhage
Symptomatic intracranial hemorrhage within 48 hours | within 48 hours after endovascular treatment
  evaluate intracranial hemorrhage (Heidelberg classification)
Mortality within 90 days | 90 days
  evaluate death rate of the two treatment groups
Procedural-related complications | within 90 days
  evaluate complications
Severe adverse events | within 90 days
  evaluate any adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Qingwu Yang, MD, Principal Investigator — Neurology, Xinqiao Hospital of the Army Medical University; Raul G Nogueira, MD, Principal Investigator — Marcus Stroke & Neuroscience Center, Grady Memorial Hospital, Emory University, Atlanta, USA; Jeffrey L Saver, MD, Principal Investigator — Neurology, University of California, Los Angeles, USA; Wenjie Zi, MD, Principal Investigator — Neurology, Xinqiao Hospital of the Army Medical University
Locations (6):
- China (6):
  - Xinqiao Hospital of Army Medical University, Chongqing, Chongqing Municipality
  - The Second Hospital of Jiaozuo, Jiaozuo, Henan
  - Wuhan No. 1 Hospital, Wuhan, Hubei
  - The First Affiliated Hospital, Hengyang Medical School, University of South China, Hengyang, Hunan
  - Xiangtan Central Hospital, Xiangtan, Hunan
  - The 904th Hospital of CPLA, Wuxi, Jiangsu

IPD SHARING:
Plan to Share IPD: Yes
study data without patient information
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Related papers published 3 months later, the IPD will be shared.
Access Criteria: yangqwmlys@163.com ziwenjie1981@163.com

REFERENCES:
- [Background] Campbell BCV, Mitchell PJ, Churilov L, Yassi N, Kleinig TJ, Dowling RJ, Yan B, Bush SJ, Thijs V, Scroop R, Simpson M, Brooks M, Asadi H, Wu TY, Shah DG, Wijeratne T, Zhao H, Alemseged F, Ng F, Bailey P, Rice H, de Villiers L, Dewey HM, Choi PMC, Brown H, Redmond K, Leggett D, Fink JN, Collecutt W, Kraemer T, Krause M, Cordato D, Field D, Ma H, O'Brien B, Clissold B, Miteff F, Clissold A, Cloud GC, Bolitho LE, Bonavia L, Bhattacharya A, Wright A, Mamun A, O'Rourke F, Worthington J, Wong AA, Levi CR, Bladin CF, Sharma G, Desmond PM, Parsons MW, Donnan GA, Davis SM; EXTEND-IA TNK Part 2 investigators. Effect of Intravenous Tenecteplase Dose on Cerebral Reperfusion Before Thrombectomy in Patients With Large Vessel Occlusion Ischemic Stroke: The EXTEND-IA TNK Part 2 Randomized Clinical Trial. JAMA. 2020 Apr 7;323(13):1257-1265. doi: 10.1001/jama.2020.1511. PMID 32078683
- [Background] Mai LM, Oczkowski W. Tenecteplase before thrombectomy for ischemic stroke improved reperfusion compared with alteplase. Ann Intern Med. 2018 Aug 21;169(4):JC20. doi: 10.7326/ACPJC-2018-169-4-020. No abstract available. PMID 30128510
- [Background] Campbell BCV, Mitchell PJ, Churilov L, Yassi N, Kleinig TJ, Dowling RJ, Yan B, Bush SJ, Dewey HM, Thijs V, Scroop R, Simpson M, Brooks M, Asadi H, Wu TY, Shah DG, Wijeratne T, Ang T, Miteff F, Levi CR, Rodrigues E, Zhao H, Salvaris P, Garcia-Esperon C, Bailey P, Rice H, de Villiers L, Brown H, Redmond K, Leggett D, Fink JN, Collecutt W, Wong AA, Muller C, Coulthard A, Mitchell K, Clouston J, Mahady K, Field D, Ma H, Phan TG, Chong W, Chandra RV, Slater LA, Krause M, Harrington TJ, Faulder KC, Steinfort BS, Bladin CF, Sharma G, Desmond PM, Parsons MW, Donnan GA, Davis SM; EXTEND-IA TNK Investigators. Tenecteplase versus Alteplase before Thrombectomy for Ischemic Stroke. N Engl J Med. 2018 Apr 26;378(17):1573-1582. doi: 10.1056/NEJMoa1716405. PMID 29694815
- [Result] Zi W, Qiu Z, Li F, Sang H, Wu D, Luo W, Liu S, Yuan J, Song J, Shi Z, Huang W, Zhang M, Liu W, Guo Z, Qiu T, Shi Q, Zhou P, Wang L, Fu X, Liu S, Yang S, Zhang S, Zhou Z, Huang X, Wang Y, Luo J, Bai Y, Zhang M, Wu Y, Zeng G, Wan Y, Wen C, Wen H, Ling W, Chen Z, Peng M, Ai Z, Guo F, Li H, Guo J, Guan H, Wang Z, Liu Y, Pu J, Wang Z, Liu H, Chen L, Huang J, Yang G, Gong Z, Shuai J, Nogueira RG, Yang Q; DEVT Trial Investigators. Effect of Endovascular Treatment Alone vs Intravenous Alteplase Plus Endovascular Treatment on Functional Independence in Patients With Acute Ischemic Stroke: The DEVT Randomized Clinical Trial. JAMA. 2021 Jan 19;325(3):234-243. doi: 10.1001/jama.2020.23523. PMID 33464335
- [Derived] Qiu Z, Li F, Sang H, Yuan G, Xie D, Zhou K, Li M, Meng Z, Kong Z, Ruan Z, Li C, Yang G, Wu J, Long C, Yang B, Hu H, Li Y, Luo J, Shi Z, Huang X, Jiang S, Yi T, Zeng G, Liu J, Luo X, Liu S, Chang M, Wu Y, Tang Y, Tian Z, Yan Z, Zhao H, Peng Y, Dai H, Zhou P, Li H, Liu W, Song D, Lei B, Xia Z, Tan X, Zhao M, Feng X, Cai L, Li Q, Wu Y, Jiang B, Tian Y, Li L, Jiang L, Long X, You F, Tao J, Zhou J, Wu D, Zheng C, Yin C, Wang D, Lu M, Albers GW, Nogueira RG, Campbell BCV, Nguyen TN, Saver JL, Zi W, Yang Q; BRIDGE-TNK Trial Investigators. Intravenous Tenecteplase before Thrombectomy in Stroke. N Engl J Med. 2025 Jul 10;393(2):139-150. doi: 10.1056/NEJMoa2503867. Epub 2025 May 21. PMID 40396577
- [Derived] Qiu Z, Li F, Xie D, Yuan G, Nguyen TN, Zhou K, Nogueira RG, Saver JL, Campbell BCV, Albers GW, Sang H, Li L, Tian Y, Meng Z, Wang D, Zi W, Yang Q; BRIDGE-TNK investigators. Efficacy and Safety of Intravenous Tenecteplase Before Endovascular Thrombectomy for Acute Ischemic Stroke: The Multicenter, Randomized, BRIDGE-TNK Trial Protocol. J Am Heart Assoc. 2024 Nov 5;13(21):e036765. doi: 10.1161/JAHA.124.036765. Epub 2024 Oct 22. PMID 39435713